CLINICAL TRIAL: NCT06157255
Title: An Open-Label, Two-Part Sequential Study Designed to Assess the Mass Balance Recovery, Absorption, Metabolism, Excretion of [14C]AZD4604 and the Absolute Bioavailability of AZD4604 in Healthy Male and Female Subjects
Brief Title: An ADME Study of [14C]AZD4604 and the Absolute Bioavailability of AZD4604
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8210C00004
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD4604 (Experimental): In Part 1, one 30 ug dose of [14C]AZD4604 Solution for Infusion 6 ug/mL (NMT 37.0 kBq/5 mL) and one 3 mg dose of AZD4604 Inhalation Powder, 1 mg (as 3 x 1 mg). In Part 2, one 4 mg dose of [14C]AZD4604 Oral Solution, 4 mg (NMT 37.0 kBq).
  Interventions: Drug: AZD4604 Inhalation Powder, 1 mg; Drug: [14C]AZD4604 Solution for Infusion 6 μg/mL (NMT 37.0 kBq/5 mL); Drug: [14C]AZD4604 Oral Solution, 4 mg (NMT 37.0 kBq)

INTERVENTIONS:
Drug: AZD4604 Inhalation Powder, 1 mg — 3 mg dose, inhaled, fasted
  Other Names: AZD4604
Drug: [14C]AZD4604 Solution for Infusion 6 μg/mL (NMT 37.0 kBq/5 mL) — 30 μg, intravenous, fasted
  Other Names: AZD4604
Drug: [14C]AZD4604 Oral Solution, 4 mg (NMT 37.0 kBq) — 4 mg, oral, fasted
  Other Names: AZD4604

SUMMARY:
The Sponsor is developing the test medicine, AZD4604, as a potential treatment for asthma. Asthma is a common lung condition caused by inflammation (swelling) of the breathing tubes that carry air in and out of the lungs, causing occasional breathing difficulties such as wheezing, shortness of breath, chest tightness and cough.

This study in healthy volunteers will explore the following questions.

* Does the test medicine cause any important side effects?
* What are the blood levels of the test medicine and how quickly does the body get rid of it?
* How much of the test medicine gets into the bloodstream?
* How does the body break down and get rid of the test medicine?

This study will take place at one non-NHS site in Nottingham, and plans to enrol 8 healthy men and women aged 18-65 years who will be involved in both parts of the study.

DETAILED DESCRIPTION:
The Sponsor is developing the test medicine, AZD4604, as a potential treatment for asthma. Asthma is a common lung condition caused by inflammation (swelling) of the breathing tubes that carry air in and out of the lungs, causing occasional breathing difficulties such as wheezing, shortness of breath, chest tightness and cough.

In this study, healthy volunteers will be given single doses of test medicine to find out how the body breaks down and gets rid of the test medicine. Two doses of the test medicine will be 'radiolabelled' - they will contain a small amount of radioactivity (Carbon-14) - so that it can be tracked in the body.

This study in healthy volunteers will explore the following questions.

* Does the test medicine cause any important side effects?
* What are the blood levels of the test medicine and how quickly does the body get rid of it?
* How much of the test medicine gets into the bloodstream?
* How does the body break down and get rid of the test medicine?

This study will take place at one non-NHS site in Nottingham.

It plans to enrol 8 healthy men and women aged 18-65 years who will be involved in both parts of the study.

In Part 1, volunteers will receive a dose of test medicine containing a very tiny amount of radio label, by injection into a vein, shortly followed by a single inhaled dose of the test medicine. In Part 2, volunteers will receive a dose of test medicine containing a very tiny amount of radio label, by mouth. In both parts volunteers will stay in the clinic for 15 nights, there will be a minimum 21 day washout period between each study part, and it will take up to 13 weeks to finish the study. A follow-up phone call will be conducted 6 to 10 days after discharge from Part 2.

Blood and urine samples will be collected to do safety tests. Over a period of at least 15 days for each part, many blood samples will be taken and volunteers will collect all their urine and faeces so that the amount of test medicine and its breakdown products can be measured.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Must be willing and able to communicate and participate in the whole study
* Healthy males or non-pregnant, non-lactating healthy female subjects aged 18 to 65 years inclusive at the time of signing informed consent
* Females must have a negative serum pregnancy test at screening and a negative urine pregnancy test on admission to the unit, must not be lactating and not intending to become pregnant during their study participation, confirmed at screening and admission/pre-dose and fulfil the criteria detailed in the Clinical Protocol
* Must agree to adhere to the contraception requirements defined in the Clinical Protocol
* Body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive and weight at least 50 kg and no more than 100 kg inclusive
* Must have regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day)
* Screening/pre-dose FEV1 >80% of the predicted value for their age, gender, height and race
* Screening/pre-dose FEV1/forced vital capacity (FVC) >0.70

Exclusion Criteria:

* History of any clinically significant disease or disorder (e.g. cardiovascular pulmonary, GI, liver, renal, neurological, musculoskeletal ,endocrine, metabolic, malignant, psychiatric, major physical impairment, skin abnormalities and glucose metabolism abnormalities) which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study
* History or presence of GI, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Subjects with a history of asymptomatic gall stones
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4604. Hay fever is allowed unless it is active
* History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or GI disease, neurological or psychiatric disorder, as judged by the investigator
* Subjects with a milk or milk protein allergy
* Subjects who have had any malignancy or neoplastic disease (except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated and considered cured)
* Subjects with history or any ongoing, chronic or recurrent infectious disease, herpes, or evidence of tuberculosis infection
* Subjects with risk factors for thrombosis or any history of thrombosis
* Subjects with a previous history of pneumonia (even if effectively treated)
* History of infantile bronchiolitis, a history of asthma, adverse reaction or allergy to the inhaled medication AZD4604 or any excipients
* Upper respiratory tract infection (excluding otitis media) within 14 days of first admission, or lower respiratory tract infection within the last 3 months
* Acute diarrhoea or constipation in the 7 days before the predicted first dosing date. If screening occurs >7 days before the first dosing date, this criterion will be determined on first dosing date. Diarrhoea will be defined as the passage of liquid faeces and/or a stool frequency of greater than 3 times per day. Constipation will be defined as a failure to open the bowels less frequently than every other day.
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis as judged by the investigator. Subjects with Gilbert's Syndrome are allowed.
* Subjects with any of the following at screening:

White blood cell count ˂3.0 × 109/L Absolute neutrophil count ˂1.8 × 109/L Lymphocyte count ˂1.0 × 109/L

* Any clinically significant abnormal findings in vital signs, at screening or pre-dose, as judged by the investigator
* Any clinically significant abnormalities on 12-lead ECG, at screening or pre-dose, as judged by the investigator
* Any positive result at screening for serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), and human immunodeficiency virus (HIV) 1 and 2 antibody
* Any positive QuantiFERON®-TB Gold test at screening
* Subjects with haemoglobin <(LLN + 1 g/dL) at screening
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <80 mL/min using the Cockcroft-Gault equation
* Has received another new chemical or biologic entity (defined as a compound which has not been approved for marketing) within the 90 days prior to the planned first dosing date, or less than 5 elimination half-lives prior to the planned first dosing date, whichever is longer. Note: subjects consented and screened, but not randomised/enrolled in this study or a previous Phase I study, are not excluded
* Subjects who report to have previously received AZD4604
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study
* Subjects who have been administered a [14C]-labelled IMP in an ADME study in the last 12 months
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening
* Use of any prescribed or non-prescribed medication including antacids, analgesics (other than up to 4 g of paracetamol/acetaminophen per day, hormonal contraception), herbal remedies, and megadose vitamins and minerals (intake of >3 times the recommended daily dose) during the two weeks prior to the first administration of IMP or longer if the medication has a long half-life Exceptions may apply, as determined by the investigator, if each of the following criteria are met: medication with a short half-life if the washout is such that no pharmacodynamic activity is expected by the time of dosing with IMP; and if the use of medication does not jeopardise the safety of the trial subject; and if the use of medication is not considered to interfere with the objectives of the study.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks or 5 half-lives, whichever is longer, prior to the first administration of IMP
* Subjects who have received any live, attenuated or mRNA vaccine within 4 weeks prior to the first administration of IMP
* Known or suspected history of alcohol or drug abuse in the past 2 years or excessive intake of alcohol (>21 units per week for men and >14 units per week for women [1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type]) or as judged by the investigator
* A confirmed positive alcohol breath test at screening or admission
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening
* A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
* Confirmed positive drugs of abuse test result at screening or admission
* Excessive intake of caffeine-containing drinks or food (e.g. coffee, tea, chocolate) as judged by the investigator. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day (e.g. >5 cups of coffee) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the investigational site.
* Male subjects with pregnant partners
* Involvement of any Astra Zeneca, Quotient or study site employee or their close relatives
* Judgment by the investigator that the volunteer should not participate in the study if they have any ongoing or recent (i.e. during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements
* Subjects who cannot communicate reliably with the Investigator.
* Vulnerable subjects, e.g. kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order
* Subjects who are unable to demonstrate effective inhalation technique with DPI at screening, Day -1 or pre-dose of Part 1 (if applicable)
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Amount of AZD4604 excreted (Ae) - Part 1 | Urine and faecal sample collection from pre-dose to 336 hours post-dose
  Mass balance of total radioactivity (TR) of [14C]AZD4604 in urine and faeces
Amount of AZD4604 excreted expressed as a fraction of dose excreted (Fe) - Part 1 | Urine and faecal sample collection from pre-dose to 336 hours post-dose
  Mass balance of total radioactivity (TR) of [14C]AZD4604 in urine and faeces
The cumulative amount of AZD4604 excreted (CumAe) - Part 1 | Urine and faecal sample collection from pre-dose to 336 hours post-dose
  Mass balance of total radioactivity (TR) of [14C]AZD4604 in urine and faeces
Cumulative amount of AZD4604 excreted expressed as a fraction of dose excreted (CumFe) - Part 1 | Urine and faecal sample collection from pre-dose to 336 hours post-dose
  Mass balance of total radioactivity (TR) of [14C]AZD4604 in urine and faeces
Time to maximum concentration (tmax) for AZD4604 and total radioactivity - Part 1 | Plasma sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 and [14C]AZD4604 in plasma
Area under the curve from time 0 extrapolated to infinity for AZD4604 and total radioactivity (AUC-inf) - Part 1 | Plasma sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 and [14C]AZD4604 in plasma
Maximum observed concentration (Cmax) for AZD4604 and total radioactivity - Part 1 | Plasma sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 and [14C]AZD4604 in plasma
Area under the curve from time 0 to the time of the last measurable concentration for AZD4604 and total radioactivity (AUC0-t) - Part 1 | Plasma sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 and [14C]AZD4604 in plasma
Area under the curve from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity (AUCextrap) and total radioactivity - Part 1 | Plasma sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 and [14C]AZD4604 in plasma
Terminal elimination half-life of AZD4604 (t1/2) and total radioactivity - Part 1 | Plasma sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 and [14C]AZD4604 in plasma
First order rate constant associated with the terminal (log-linear) portion of the curve for AZD4604 (λz) and total radioactivity - Part 1 | Plasma sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 and [14C]AZD4604 in plasma
Total body clearance calculated after a single IV administration (CL) - Part 1 | Plasma sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 and [14C]AZD4604 in plasma
Total body clearance calculated after a single extravascular administration where F (fraction of dose bioavailable) is unknown (CL/F) - Part 1 | Plasma sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 and [14C]AZD4604 in plasma
Volume of distribution based on the terminal phase calculated using AUC(0-inf) after a single IV administration (Vz) - Part 1 | Plasma sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 and [14C]AZD4604 in plasma
Volume of distribution based on the terminal phase calculated using AUC(0-inf) after a single extravascular administration where F (fraction of dose bioavailable) is unknown (Vz/F) - Part 1 | Plasma sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 and [14C]AZD4604 in plasma
Assessment of metabolites in plasma, urine and faeces by liquid chromatography-radiochemical-detection and subsequent mass spectrometry - Part 1 | Plasma, urine and faces sample collection from pre-dose to 336 hours post-dose
  Metabolite profiling and structural identification from plasma, urine and faecal samples
Amount of AZD4604 excreted (Ae) - Part 2 | Urine and faecal sample collection from pre-dose to 336 hours post-dose
  Mass balance of total radioactivity (TR) of [14C]AZD4604 in urine and faeces
Amount of AZD4604 excreted expressed as a fraction of dose excreted (Fe) - Part 2 | Urine and faecal sample collection from pre-dose to 336 hours post-dose
  Mass balance of total radioactivity (TR) of [14C]AZD4604 in urine and faeces
The cumulative amount of AZD4604 excreted (CumAe) - Part 2 | Urine and faecal sample collection from pre-dose to 336 hours post-dose
  Mass balance of total radioactivity (TR) of [14C]AZD4604 in urine and faeces
Cumulative amount of AZD4604 excreted expressed as a fraction of dose excreted (CumFe) - Part 2 | Urine and faecal sample collection from pre-dose to 336 hours post-dose
  Mass balance of total radioactivity (TR) of [14C]AZD4604 in urine and faeces
Time to maximum concentration (tmax) for AZD4604 and total radioactivity - Part 2 | Plasma and whole blood sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 in plasma and whole blood
Area under the curve from time 0 extrapolated to infinity for AZD4604 and total radioactivity (AUC-inf) - Part 2 | Plasma and whole blood sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 in plasma and whole blood
Maximum observed concentration (Cmax) for AZD4604 and total radioactivity - Part 2 | Plasma and whole blood sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 in plasma and whole blood
Area under the curve from time 0 to the time of the last measurable concentration for AZD4604 and total radioactivity (AUC0-t) - Part 2 | Plasma and whole blood sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 in plasma and whole blood
Area under the curve from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity (AUCextrap) and total radioactivity - Part 2 | Plasma and whole blood sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 in plasma and whole blood
Terminal elimination half-life of AZD4604 (t1/2) and total radioactivity - Part 2 | Plasma and whole blood sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 in plasma and whole blood
First order rate constant associated with the terminal (log-linear) portion of the curve for AZD4604 (λz) and total radioactivity - Part 2 | Plasma and whole blood sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 in plasma and whole blood
Total body clearance calculated after a single extravascular administration where F (fraction of dose bioavailable) is unknown (CL/F) - Part 2 | Plasma and whole blood sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 in plasma and whole blood
Volume of distribution based on the terminal phase calculated using AUC(0-inf) after a single extravascular administration where F (fraction of dose bioavailable) is unknown (Vz/F) - Part 2 | Plasma and whole blood sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 in plasma and whole blood
Renal clearance calculated using plasma AUC of AZD4604 and total radioactivity - Part 2 | Plasma and whole blood sample collection from pre-dose to 336 hours post-dose
  PK of AZD4604 in plasma and whole blood
Assessment of metabolites in plasma, urine and faeces by liquid chromatography-radiochemical-detection and subsequent mass spectrometry - Part 2 | Plasma, urine and faces sample collection from pre-dose to 336 hours post-dose
  Metabolite profiling and structural identification from plasma, urine and faecal samples

SECONDARY OUTCOMES:
Absolute bioavailability - Part 1 | Plasma sample collection from pre-dose to 336 hours post-dose
  Absolute bioavailability (Finh) based on AUC0-inf of inhaled administration compared to IV administration, adjusted for dose
Identification of the chemical structure of each metabolite accounting for more than 10% by AUC of circulating TR and/or accounting for 10% or more of the dose in excreta | Urine and faecal sample collection from pre-dose to 336 hours post-dose
  Identification of chemical structure of each metabolite accounting for more than 10% of circulating TR or accounting for 10% more of the dose in urine and faeces
Number of subjects with treatment-related adverse events - Part 1 and Part 2 | Through study duration, approximately 13 weeks
  To provide additional safety and tolerability information for AZD4604 by assessing the incidence of AEs
Blood:plasma concentration ratios - Part 2 | Whole blood samples and plasma samples collected from pre-dose until 336 hours post-dose
  Blood:plasma concentration ratios of total radioactivity
Absolute bioavailability - Part 2 | Plasma sample collection from pre-dose to 336 hours post-dose
  Absolute bioavailability (Finh) based on AUC0-inf of oral administration compared to IV administration, adjusted for dose

CONTACTS AND LOCATIONS:
Overall Officials: Somasekhara Menakuru, MBBS, MS, MRCS, DPM, MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Research Site, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to teh EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-levels data in an approved sponsors tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the disclosure statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-DT.pharmacm.com/DT/Home